CLINICAL TRIAL: NCT02208752
Title: The Effect of a Pre-operative Exercise Program on Pain and Function in Patients With Full Thickness Rotator Cuff Tear Waiting for Surgical Repair.
Brief Title: The Effect of a Pre-operative Exercise Program for Patients With Full Thickness Rotator Cuff Tear Waiting for Surgical Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, François Desmeules, Principal researcher, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CARM2014
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff tears; ultrasound measure; pain; range of motion; muscle force
MeSH Terms: conditions — Rotator Cuff Injuries; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercises (Active Comparator): exericises on motor control and strengthening exercises on the Rotator Cuff
  Interventions: Other: Exercises
- Control group- No exercises (Placebo Comparator): No exercises
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — exercise program on strengthening the rotator cuff muscles and motor control of the scapula

SUMMARY:
This is a randomised controlled study involving a group of 20 patients- 10 patients in a control group, 10 patients in treatment group. The treatment group consists of exercises with theraband for the shoulder and exercises of motor control of the scapula. The purpose of the study is to measure the effects of a pre-operative physiotherapy program for patients awaitng for rotator cuff surgery, The duration of the pilot project is 4 weeks.

DETAILED DESCRIPTION:
This study is taken place in a genral hospital using the waiting list in the orthopedic surgery department- only patients awaitng for rotator cuff surgery are included. a randomised process of a block will be used. There will be 2 groups of patients an active comparator and no intervention. All patients at the beginning of the project and after 4 weks will have an evaluation on range of motion, strength, acromial humeral mesurement done by ultrasound and questionnaire on pain(DASH) and quality of life( WORC). At 8 weeks all patients will fill in the 2 questionnaires on DASH and WORC.

ELIGIBILITY:
Inclusion Criteria:

* Patients waitng for surgery at Cite de la Sante Hospital

Exclusion Criteria:

* Glenohumeral Arthirtis
* Shoulder fracture
* Corticosteriod injections
* Rupture of rotator cuff tear of more than 3 cm
* CSST- Workman's compensation
* Central and peripheral neuropathy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
WORC questionnaire | 30 days
  To evaluate function and quality of life at 0 weeks and 4 weeks

SECONDARY OUTCOMES:
DASH questionnaire | 30 days
  To evaluate pain at 0 weeks and 4 weeks
Ultrasound measures | 30 days
  Mesurement distance of acromial-humerale distance at 0 and 4 weeks
range of motion | 30 days
  measurement of joint movement (active and passif range of motion) with goniometer at 0 and 4 week
strength | 30 days
  measurement of isometric strength with the Nicolas dynamometer at 0 week and 4 week.

CONTACTS AND LOCATIONS:
Overall Officials: François Desmeules, Phd, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital Cite-de-la-Santé, Laval, Quebec, Canada